CLINICAL TRIAL: NCT03175861
Title: Multiscale Modeling / Simulation of the Response to Pulmonary Stereotactic Hypofractionated Irradiation
Brief Title: Modeling of the Response to Hypofractionated Stereotactic Pulmonary Irradiation
Acronym: MUMOFRAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: MUMOFRAT
Record Dates: First submitted 2017-05-23; First posted 2017-06-05 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Stereotactic radiotherapy — The patient will have an initial pre-therapeutic assessment in the 8 weeks before the start of radiotherapy Then, radiation therapy planning with 3 free breathing 4D (4 dimensions) scanners performed over 8 days without injection of iodinated contrast agent.
  Then the patient will receive his treatment by conventional stereotactic radiotherapy

SUMMARY:
Identify 18-Fluorodeoxyglucose (18F-FDG) positron emission tomography-computed tomography (PET-CT) parameters predictive of tumor response and local control

DETAILED DESCRIPTION:
The identification of robust prognostic and predictive markers could allow the individualization of pulmonary stereotactic radiotherapy treatments and the selection of patients at high risk of relapse, who could then benefit from a dose escalation in order to increase the chances of local control .

Beyond the pulmonary RTS (Radiotherapy in stereotactic condition), this study will aim to generate one or more models of multi-scale response to hypofractionated irradiation from biomarkers (biological or images) extracted from preclinical or clinical literature data and to allow simulations of Various modified fractionation irradiation schemes, potentially leading to new regimens that reduce side effects and increase therapeutic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Performance Index WHO (World Health Organization) ≤ 2
* Bronchopulmonary carcinoma not in small cells proved histologically or cytologically (epidermoid, adenocarcinoma, or large cell carcinoma).
* Tumor classified T1 - T2 (Tumor=1-2) N0 (Node=0) M0 (Metastasis=0) and diameter ≤ 5 cm or Tumor classified T3 (≤5cm) N0M0 of the chest wall
* Tumor located more than 2 cm from the trachea and bronchus stem and more than 1.5 cm from the organs at risk
* Medically inoperable or refusing surgery
* Indication of stereotactic radiotherapy validated in multidisciplinary consultation meeting
* Formulation of consent

Exclusion Criteria:

* Age <18 years.
* History of pulmonary irradiation
* Pulmonary surgery of the tumor
* Different histology of non-small cell carcinoma
* Patient with a T2 or T3> 5 cm tumor or patients with a T3 tumor invading a structure other than the chest wall
* Patient with a tumor within 2 cm of the trachea and bronchus stem and within 1.5 cm of the organs at risk in the proximal area of the no fly zone (defined as a volume Located 2 cm in all directions of the proximal bronchial tree - Pulmonary metastases
* Declared pregnancy, breast-feeding
* Refusal to use effective contraception
* Against indication to the realization of the PET to the 18FDG (18-fluorodeoxyglucose)(uncontrolled diabetes)
* Refusal or inability to consent to participate in the study.
* Estimated life expectancy <2 months in the absence of treatment
* Other invasive tumors diagnosed in the previous 2 years, with the exception of non-melanocytic cutaneous carcinomas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All major patients requiring stereotactic radiotherapy for non-small cell bronchopulmonary carcinoma.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Kinetics of PET-CT parameters : standardized uptake value (SUV) max | 2 years
  SUV max will be measured before and after stereotactic irradiation.
Tumor metabolic response | 2 years
  Tumor metabolic response, as assessed on 18F-FDG PET-CT at 6 months of end of radiotherapy
Local control | 2 years
  Local control defined by the absence of progression in the irradiated area
Kinetics of PET-CT parameters : metabolic tumor volume | 2 years
  Metabolic tumor volume (MTV) will be measured before and after stereotactic irradiation.
Kinetics of PET-CT parameters : texture parameters :quantitative extraction of images by specific software | 2 years
  The first-order form parameters and statistical parameters, the second order (based on the matrix of co-occurrence of the grey levels and the matrix of differences of grey levels) and of the third order (based on the matrices of alignment of the grey levels and the matrices of sizes of zones) will be studied.

SECONDARY OUTCOMES:
Kinetics of serum markers | 2 years
  The kinectic will be measured
Predictive power of serum markers for tumor response and local control | 2 years
  This predictive power will be measured
Predictive power of metabolic imaging parameters for tumor response and local control Predictive power of metabolic imaging parameters for tumor response and local control | 2 years
  This predictive power will be measured
Correlation between these parameters | 2 years
  The correlation will be measured
Survival in disease | 2 years
  The survival in desease will be observed
Survival without metastasis at a distance | 2 years
  The survival without metastasis will be observed
Radiation-induced toxicity | 2 years
  The radiation-induced toxicity will be observed

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Schick, Doctor, Principal Investigator — University Hospital, Brest
Locations (4):
- France (4):
  - CHRU de Brest, Brest
  - Centre Eugène Marquis, Rennes
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Clinique d'Oncologie et Radiothérapie, Tours